CLINICAL TRIAL: NCT01048346
Title: Efficacy of the Individual Placement and Support (IPS) Model for Consumers With Disability and Substance Use Disorders
Brief Title: Efficacy of the Individual Placement and Support (IPS) Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Substance Use Disorders
Keywords: employment, disabilities
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- supported employment (Experimental): Study consists of one experimental group and one control group. The intervention group received IPS
  Interventions: Behavioral: Individual Placement and Support Model

INTERVENTIONS:
Behavioral: Individual Placement and Support Model — Psychosocial intervention involving an employment specialist working with participants recruited into the study and assisting with employment.
  Other Names: Supported employment intervention

SUMMARY:
Hypothesis 1. Consumers with disabilities and co-occurring SUD receiving IPS will be more likely to be competitively employed (defined as 1 or more days of work over the past 30 days) at 3, 6 and 12 months following the initiation of vocational treatment goals when compared to a group receiving standard services.

Hypothesis 2. Consumers with disabilities and co-occurring SUD receiving IPS when compared to the comparison group will 1.) be more successful in achieving their employment goals as indicated by the ratio of hours worked to desired hours worked; 2.) become competitively employed sooner; 3.) earn higher wages, 4.) have greater job satisfaction, 5.) have greater economic satisfaction; 6.) have greater life satisfaction, 7.) have greater self-esteem, and 8.) have fewer days of using substances during follow-up points.

DETAILED DESCRIPTION:
Hypothesis 1. Consumers with disabilities and co-occurring SUD receiving IPS will be more likely to be competitively employed (defined as 1 or more days of work over the past 30 days) at 3, 6 and 12 months following the initiation of vocational treatment goals when compared to a group receiving standard services.

Hypothesis 2. Consumers with disabilities and co-occurring SUD receiving IPS when compared to the comparison group will 1.) be more successful in achieving their employment goals as indicated by the ratio of hours worked to desired hours worked; 2.) become competitively employed sooner; 3.) earn higher wages, 4.) have greater job satisfaction, 5.) have greater economic satisfaction; 6.) have greater life satisfaction, 7.) have greater self-esteem, and 8.) have fewer days of using substances during follow-up points.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes consumers who are between the ages of 18-65, able to provide informed consent for participation, and are initiating an employment goal in their treatment plan.

Exclusion Criteria:

* Exclusion criteria includes anyone who is currently employed and has been for the past 30 days, have an open case with the Ohio Rehabilitation Services Commission, or have an open case with another vocational rehabilitation provider.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2009-05-01 (Actual)

PRIMARY OUTCOMES:
Competitive employment | May 2005 - May 2009

SECONDARY OUTCOMES:
life satisfaction, job satisfaction, self-esteem, substance and alcohol use | May 2005 - May 2009

CONTACTS AND LOCATIONS:
Locations (1):
- CAM, Dayton, Ohio, United States